CLINICAL TRIAL: NCT03690609
Title: CytoQuel: Clinical Documentation on Effects on Chronic Pain, Wellness, and Reduction of Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Research director, Natural Immune Systems Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NIS143002
Record Dates: First submitted 2018-09-06; First posted 2018-10-01 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceutical intervention, 3 capsules daily. (Active Comparator): Participants will consume the nutraceutical blend CytoQuel at a dose of 1850 mg, by consuming 3 capsules daily in the morning.
  Interventions: Dietary Supplement: CytoQuel
- Nutraceutical intervention, 2 capsules twice daily. (Active Comparator): Participants will consume the nutraceutical blend CytoQuel at a dose of 1850 mg, by consuming 4 capsules daily: Two in the morning and two later in the day.
  Interventions: Dietary Supplement: CytoQuel

INTERVENTIONS:
Dietary Supplement: CytoQuel — 3 capsules daily.
  Arms: Nutraceutical intervention, 3 capsules daily.
Dietary Supplement: CytoQuel — 2 capsules twice daily.
  Arms: Nutraceutical intervention, 2 capsules twice daily.

SUMMARY:
The purpose for this protocol is to perform an open-label parallel-arm clinical study in healthy subjects to evaluate the efficacy of a nutraceutical product on chronic pain, vascular health, inflammation, and overall wellness.

DETAILED DESCRIPTION:
This is an open-label proof-of-concept human clinical study on the effects of consumption of a nutraceutical blend. Data collection will include a core set of data pertaining to chronic pain and inflammatory markers. Additional data collection will include blood pressure, weight, and overall wellness.

An open-label study design will be used to evaluate the effects of consumption of the nutraceutical product CytoQuel. The product is marketed broadly for many types of inflammation-related health issues. The study is of 8 weeks' duration, with evaluation at baseline, 2, and 8 weeks of product consumption. Study participants will be randomized to one of two groups, taking either 3 caps once daily, or two caps twice daily.

At each visit, the following measurements and procedures are performed: Blood pressure and ankle brachial index, questionnaires pertaining to pain and activities of daily living, and a blood draw. The blood is used for testing of cytokines and vascular health related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adult people of either gender;
* Age 30-75 years (inclusive);
* BMI between 20.0 and 34.9 (inclusive);
* Experiencing chronic pain in at least one specific anatomical area for more than 6 months.

Exclusion Criteria:

* Active uncontrolled auto-immune disease (for example: rheumatoid arthritis, lupus, inflammatory bowel disease, Celiac disease);
* Known active cardiovascular health issues;
* Cancer during past 12 months;
* Chemotherapy during past 12 months;
* Currently taking blood pressure medication;
* Currently taking blood thinning medication (81mg aspirin allowed);
* Currently taking cholesterol-lowering medication (for example: statins);
* Currently taking Coumadin;
* Currently taking nutritional supplements judged by the study coordinator to negate or camouflage the effects of the test product;
* Currently taking prescription pain medications;
* Getting regular joint injections (such as cortisone shots);
* Major surgery within the past 3 months;
* Major trauma within the past 3 months;
* Any other condition or observation that the investigator judges may adversely affect the person's ability to complete the study;
* Any other significant disease or disorder that the investigator judges may put the subject at risk because of participation in the study, or may influence the result of the study;
* Hypersensitivity or known allergy to green tea or black tea;
* Participation in another research study involving an investigational product in the past month;
* Planned surgery within 2 weeks of completing the study;
* Previous major surgery to stomach or intestines [(absorption of test product may be altered) minor surgery is not a problem, including appendix and gallbladder removal];
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Women who are pregnant, nursing, or trying to become pregnant.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Change in pain level from baseline | 8 weeks.
  Pain questionnaire: Scale 0-10, with 0 being pain-free and 10 being the most pain. Change from baseline will be evaluated.

SECONDARY OUTCOMES:
Change in blood pressure from baseline | 8 weeks.
  Systolic and diastolic blood pressure.

OTHER OUTCOMES:
Change in Fibrinogen level from baseline | 8 weeks.
  Plasma fibrinogen level pg/mL
Change in von Willebrand Factor from baseline | 8 weeks.
  von Willebrand Factor level pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be published. At this time it is not determined whether individual data will be made available to other researchers.